CLINICAL TRIAL: NCT06896305
Title: Impact of Diet on the Effectiveness of Anti-TNF Therapy in Inflammatory Bowel Disease: a Prospective, Randomized, Double Arm, Open-label Study
Brief Title: Impact of Exclusion Diet in Addition to Anti-TNF Therapy in Crohn's Disease and Ulcerative Colitis: a Prospective, Randomized, Double-arm, Open-label Study
Acronym: IDEA-TNF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Tommaso Lorenzo Parigi, Gastroenterologist, IRCCS Ospedale San Raffaele
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IDEA-TNF
Record Dates: First submitted 2025-02-02; First posted 2025-03-26 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Ulcerative Colitis (UC); Crohn Disease (CD)
Keywords: Inflammatory Bowel Disease; Anti-TNF; Crohn's Disease Exclusion Diet; Ulcerative colitis; Crohn
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease; Inflammatory Bowel Diseases

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into two groups: those receiving anti-TNF treatment and dietary advice, and those receiving anti-TNF treatment only. The nature of the procedure (dietary advice) prevents the investigator and participant from being blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Patients who accept participation and are randomized to receive dietary advice on the CDED diet will be included in the intervention group.
  Interventions: Combination Product: CDED (Crohn's Disease Exclusion Diet) in addition to anti-TNF therapy
- Control group (Active Comparator): The control group will receive only anti-TNF therapy as per the standard of care and guidelines recommendation
  Interventions: Drug: Anti-TNF Therapy

INTERVENTIONS:
Combination Product: CDED (Crohn's Disease Exclusion Diet) in addition to anti-TNF therapy — Patients in the experimental group will receive professional dietary advice on how to adhere to CDED for 12 weeks, in addition to anti-TNF therapy while patients in the control group will receive only anti-TNF therapy for the entire duration of the study.
  Diet adherence is completely voluntary and is not enforced in any way. CDED is divided into 3 phases, the first two, grouped as the induction phase, with 6 weeks of strict diet and 6 weeks to gradual food reintroduction, followed by 12 weeks of patients follow-up.
  Five foods (chicken, eggs, potatoes, apple and bananas) are permitted at the start of the diet; the patient can then choose to consume a range of permitted foods at will, the variability of which increases after the first six weeks
  Arms: Intervention group
Drug: Anti-TNF Therapy — The control group will receive only anti-TNF therapy as per standard of care. This therapy is recommended by guidelines and is the cornerstone of treatment of Crohn's disease and ulcerative colitis.
  Arms: Control group

SUMMARY:
This clinical study protocol aims to prospectively compare the efficacy of standard therapy with anti-TNF agents combined with the Crohn's Disease Exclusion Diet (CDED) versus anti-TNF therapy alone in adult patients with active Crohn's disease or ulcerative colitis.

The study will involve patients starting therapy with anti-TNF agents due to active Crohn's disease or ulcerative colitis as per standard clinical practice and in accordance with European (ECCO) guidelines.

One group will receive standard medical therapy only, the other will additionally receive dietary advice on how to adhere on a specific exclusion diet, the CDED.

By prospectively evaluating the impact of this combined approach, the study seeks to provide evidence on whether CDED can improve response to treatment and therefore improve quality of life for patients with Crohn's disease and ulcerative colitis.

DETAILED DESCRIPTION:
This is a prospective interventional, single-center, double-group, open-label study.

Primary objective is to compare the efficacy of CDED in addition to anti-TNF therapy in active CD and UC versus anti-TNF therapy alone.

Secondary objective are:

* Endoscopic response
* Endoscopic remission
* Early and late efficacy and persistence of benefits
* Biochemical response
* Sonographic improvement
* Tolerability and compliance to the Crohn's Disease ExclusionDiet (CDED)
* Quality of life-Safety of the combination of biological therapy and CDED. The subjects considered are adult patients diagnosed with moderate-to-severe Crohn's disease or moderate-to-severe ulcerative colitis who are starting therapy with an approved anti-TNF agent (infliximab and adalimumab for both UC and CD, and golimumab only for UC).

ELIGIBILITY:
Inclusion Criteria:

1. Participant is willing and able to give informed consent forparticipation in the study
2. Males or Females, Adults aged 18 years or older
3. Confirmed diagnosis of moderate-to-severe Crohn's disease orulcerative colitis
4. Patients who are planned to start anti-TNF therapy
5. Ability and willingness to comply with the Crohn's DiseaseExclusion Diet (CDED)

Exclusion Criteria:

1. Patients with undetermined inflammatory bowel disease
2. Patients with metabolic or gastrointestinal conditions that couldinterfere or are incompatible with the study intervention (e.i.celiac disease, diabetes etc)
3. Patients with a body-mass index lower than 17 or greater than30
4. Patients who previously underwent intestinal resectionirrespective of cause
5. Patients currently on exclusive enteral nutrition (EEN)
6. Patients who have previously used or are currently adhering toCDED
7. Pregnant or breastfeeding women
8. Patients with a history of severe allergic reactions orintolerance to any food recommended in CDED
9. Patients with significant comorbidities that may interfere withthe study or pose a risk to the participant
10. Inability or unwillingness to comply with study protocols orfollow-up schedules

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-05-22 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of CDED in addition to anti-TNF therapy in active CD and UC versus anti-TNF therapy | Week 14/16
  Rate of symptomatic remission (Harvey - Bradshaw Index <5 for CD or Partial Mayo Score <2) for UC

SECONDARY OUTCOMES:
Endoscopic response and endoscopic remission | Week 24
  * Rate of endoscopic response for CD (SES-CD score reduction of 25% or more and of 50% or more from baseline) and for UC (endoscopic Mayo score reduction of at least 1 or more points)
  * Rate of endoscopic remission for CD (SES-CD score ≤3) and for UC (Mayo endoscopic score ≤1)
Early and late efficacy and persistence of benefits | Week 6/ Week 24
  Rate of symptomatic remission (Harvey- Bradshaw Index < 5 and Partial Mayo Score <2) at week 6 and 24
Biochemical response | Week 6, 14/16, 24
  * Change in C-reactive protein (CRP) levels from baseline
  * Change in fecal calprotectin levels from baseline
Sonographic improvement | Week 6, 14/16, 24
  * Change in BUSS (for CD) or MUC (for UC) from baseline
  * Rate of patients in transmural response (bowel wall thickness ≤3mm and no increase in bowel wall flow)
Tolerability and compliance to the Crohn's Disease Exclusion Diet (CDED) | Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12
  Percentage of patients self-reporting adherence to CDED
Quality of life assessed using the Short-IBD-Q questionnaire | Week 14/16, week 24
  Change in Short-IBDQ questionnare score. Quality of life will be assessed using the validated Italian translation of the Short-IBD-Q questionnaire
Safety of the combination of biological therapy and CDED | From baseline until the end of the study
  Incidence and type of adverse events during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Tommaso Lorenzo Parigi, MD, Principal Investigator — IRCCS Ospedale San Raffaele
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Michigan, Italy

IPD SHARING:
Plan to Share IPD: No